CLINICAL TRIAL: NCT02665039
Title: A Multicenter, Randomized Phase II Trial of Vinflunine/Gemcitabine vs Carboplatin/Gemcitabine as First Line Treatment in Patients With Metastatic Urothelial Carcinoma Unfit for Cisplatin Based Chemotherapy Due to Impaired Renal Function.
Brief Title: A Trial With Vinflunine in Patients With Metastatic Bladder Cancer and Impaired Renal Function
Acronym: VINGEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Anders Ullén (Other)
Responsible Party: Sponsor-Investigator, Dr Anders Ullén, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUCOG I
Record Dates: First submitted 2016-01-18; First posted 2016-01-27 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Renal Pelvis Cancer; Ureter Cancer; Urethra Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — vinflunine; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vinflunine + gemcitabine (Experimental): Vinflunine will be given intravenously once every 21 days, starting at a dose of:
  * 280 mg/m2 in patients with GFR 40-60 ml/min
  * 250 mg/m2 in patients aged >80 years and/or GFR 30-40 ml/min
  Gemcitabine will be given intravenously on day 1 and day 8 of every 21 day cycle, starting at a dose of 1000 mg/m2
  Interventions: Drug: Vinflunine; Drug: Gemcitabine
- Carboplatin + gemcitabine (Active Comparator): Carboplatin will be given intravenously once every 21 days, starting at a dose of AUC 4.5
  Gemcitabine will be given intravenously on day 1 and day 8 of every 21 day cycle, starting at a dose of 1000 mg/m2
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Vinflunine — Vinflunine will be given intravenously once every 21 days, starting at a dose of:
  * 280 mg/m2 in patients with GFR 40-60 ml/min
  * 250 mg/m2 in patients aged >80 years and/or GFR 30-40 ml/min
  Other Names: Javlor®
  Arms: Vinflunine + gemcitabine
Drug: Gemcitabine — Gemcitabine will be given intravenously on day 1 and day 8 of every 21 day cycle, starting at a dose of 1000 mg/m2
  Other Names: Gemzar
Drug: Carboplatin — Carboplatin will be given intravenously once every 21 days, starting at a dose of AUC 4.5
  Other Names: Karboplatin
  Arms: Carboplatin + gemcitabine

SUMMARY:
This study aim to compare the efficacy, safety and quality of life of vinflunine/gemcitabine and carboplatin/gemcitabine in patients with metastatic urothelial cancer and impaired renal function.

DETAILED DESCRIPTION:
Rational The standard first line treatment for patients with metastatic urothelial carcinoma unfit for cisplatin due to renal impairment is carboplatin containing chemotherapy, with a median overall survival of approximately 8-10 month. New, more effective regimens in terms of tumor control and quality of life are urgently needed. Vinflunine has proven efficacy in urothelial carcinoma and is registered as second line treatment. The combination of gemcitabine and vinflunine has not yet been evaluated in first line treatment for patients with metastatic urothelial carcinoma.

Objectives

* To compare the progression free survival (FPS) of vinflunine/gemcitabine versus carboplatin/gemcitabine in patients with locally advanced or metastatic transitional cell carcinoma of the urothelial tract unfit for cisplatin based chemotherapy due to impaired renal function.
* To evaluate the tumour response (ORR), overall survival (OS) and disease control rate (DCR) of vinflunine/gemcitabine versus carboplatin/gemcitabine
* To assess the safety and toxicity of vinflunine/gemcitabine versus carboplatin/gemcitabine.
* To investigate and compare Quality of life during treatment with vinflunine/gemcitabine and carboplatin/gemcitabine respectively.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent.
* Histological or cytological confirmed transitional cell carcinoma of the urothelial tract (mixed histology including transitional cell carcinoma are allowed).
* Non-curable unresectable (T4b), locally advanced (lymph node positive (N+)) or metastatic (M1) urothelial carcinoma (including renal pelvic tumours, ureteral tumours, urinary bladder tumours and urethral primary tumours).
* No prior antineoplastic chemotherapy or other anti-cancer drugs. Patients who have received neoadjuvant or adjuvant platinum containing chemotherapy and who are diagnosed with loco regional recurrent or metastatic disease after 6 months are eligible.
* Creatinine clearance 30 - 60 ml/min (measured by Iohexol or Cr-EDTA technique)
* ECOG/WHO Performance Status (PS) 0-1.

  •≥ 4 weeks since prior major surgery, ≥ 2 weeks since prior minor surgery (i.e. TUR-B) and ≥ 1 week since prior radiation therapy.
* Measurable and/or non-measurable disease using the RECIST v 1:1 criteria defined as:

  * Measurable disease: lesions that can be measured in at least one dimension and which have not been previously irradiated. Longest diameter ≥10 mm or lymph nodes ≥15 mm in short axis with CT scan or MRI.
  * Non-measurable disease: lesions which have not been previously irradiated, longest diameter <10 mm or lymph nodes 10-14 mm in short axis with CT scan or MRI, or truly non measurable lesions including bone lesions, ascites, pleural/pericardial effusion, and lymphangitis cutis/pulmonitis.
* CNS metastases and/or leptomeningeal metastases are allowed provided these have been adequately treated with radiotherapy, are stable and not generating any related neurological symptoms.
* Spinal cord compression due to metastatic lesions is allowed provided adequate surgery and/or radiotherapy has been delivered, the metastases are stable and not generating any related neurological symptoms.
* No known or suspected allergy to the investigational agents or any agents given in association with this trial.
* 18 years of age or older.
* Fertile men and women of childbearing potential must use secure contraception (women - intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), men - condom and for a female partner as described above) from before 2 months entering the study until 6 months after end of chemotherapy.

Exclusion Criteria

* Not fulfilling inclusion criteria as described above
* Pure non-transitional cell carcinoma of the urothelial.
* Pronounced hematuria in need of repeated blood transfusions, palliative radiotherapy to the bladder or palliative resection (TUR-B).
* Impaired bone marrow function defined as WBC < 3.0 x 109/L, neutrophils < 1.5 x 109/L, platelets < 125 x 109/L, haemoglobin < 100 g/L.
* Impaired liver function defined as serum bilirubin > 1.5 x upper limit of normal (ULN) and/or ASAT/ALAT > 2.5 x ULN (> 5 x ULN if known liver metastasis).
* Electrocardiogram (ECG) with significant modifications suggesting a high risk of occurrence of angina pectoris or high risk of arrhythmia.
* Other malignancies, except adequately treated basal carcinoma or squamous cell carcinoma of the skin or in-situ cervix carcinoma or incidental prostate cancer (T1a, Gleason score ≤ 6, PSA < 0.5 ng/ml), or any other tumour with a disease free survival of ≥ 5 years.
* History of serious or concurrent illness or uncontrolled medical disorder; any medical condition that might be aggravated by chemotherapy treatment or which could not be controlled; including, but not restricted to:

  * Active infection requiring antibiotics within 2 weeks before the study inclusion,
  * Unstable diabetes mellitus,
  * Hypercalcaemia >2.9 mmol/L (grade ≥ 2 according to CTCAE v 4.0),
  * Concurrent congestive heart failure NYHA (class III-IV),
  * Unstable angina pectoris, or myocardial infarction within 6 months and/or poorly controlled hypertension,
  * QTc > 450 ms at baseline,
  * Inflammatory bowel disease,
  * Peripheral neuropathy grade ≥ 2 according to CTCAE v 4.0,
* Patients who require treatment with ketoconazole, fluconazole, itraconazole, ritonavir, amprenavir, indinavir, rifampicin (any potent CYP3A4 inhibitor or inducer) or phenytoin.
* Pregnant or lactating women.
* Any psychological, familial, sociological, or geographical condition which does not permit protocol compliance and medical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization through study completion, on average within 9 months
  Defined as the duration from randomization to either confirmed progression (by RECIST) or death from any cause.

SECONDARY OUTCOMES:
Overall response rate (ORR = CR + PR) | From randomization through study completion, on average within 9 months
  Defined as best confirmed response according to RECIST through study completion from randomization to either confirmed progression (by RECIST) or death from any cause
Overall survival (OS) | From randomization to death from any cause, on average within 18 months
  Defined as the duration from randomization to death from any cause or last follow-up.
Disease control rate, DCR (=CR + PR + SD) | From randomization through study completion, on average within 9 months
  Defined as the percentage of patients who have achieved complete response, partial response and stable disease according to RECIST through study completion from randomization to either confirmed progression (by RECIST) or death from any cause
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | From the date the informed consent is signed up to 30 days after the last dose
  Treatment-related adverse events will be assessed by CTCAE v4.0. The safety profile and tolerability of vinflunine + gemcitabine compared to carboplatin + gemcitabine will be determined from the number of Adverse Events reported.
Quality of Life (QoL) assessed by QLQ-C30 | From the date the informed consent is signed up to 30 days after the last dose
  Quality of Life will be assessed by the EORTC Quality of Life Questionnaire C30 (QLQ-C30) Version 3.0. The QoL for patients treated with vinflunine + gemcitabine will be compared to patients treated with carboplatin + gemcitabine

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ullén, M.D., Ph.D., Principal Investigator — Karolinska University Hospital
Locations (2):
- Department of Oncology, Rigshospitalet, Copenhagen, Denmark
- Department of Oncology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmsten K, Jensen NV, Mouritsen LS, Jonsson E, Mellnert C, Agerbaek M, Nilsson C, Moe M, Carus A, Ofverholm E, Lahdenpera O, Brandberg Y, Johansson H, Hellstrom M, Maase HV, Pappot H, Ullen A. Vinflunine/gemcitabine versus carboplatin/gemcitabine as first-line treatment in cisplatin-ineligible patients with advanced urothelial carcinoma: A randomised phase II trial (VINGEM). Eur J Cancer. 2020 Mar;127:173-182. doi: 10.1016/j.ejca.2019.08.033. Epub 2019 Oct 22. PMID 31648851